CLINICAL TRIAL: NCT07131592
Title: The Effect of Tranexamic Acid on Drainage Volume and Time to Drain Removal in Reduction Mammaplasty Patients
Brief Title: Effect of Intravenous and Topical Tranexamic Acid on Drain Output in Breast Reduction Surgery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Katherine Carruthers, MD, MS, Primary Investigator, Assistant Professor, Division of Plastic and Reconstructive Surgery, Department of Surgery, Massachusetts General Hospital and Harvard Medical School, Boston, MA, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025P001908
Record Dates: First submitted 2025-08-05; First posted 2025-08-20 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Drain Output After Breast Reduction Surgery; Breast Reductions
Keywords: TXA; Tranexamic Acid; Breast Reduction; Postoperative Drainaige; Plastic Surgery; Randomized Controlled Trial; RCT
MeSH Terms: interventions — Tranexamic Acid; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Participants are randomized to either receive intravenous tranexamic acid (TXA) or no TXA during bilateral breast reduction surgery. Within each participant, a split-breast design is applied: one breast is treated with topical TXA through the surgical drain, while the contralateral breast receives saline
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- IV TXA + Topical TXA (Experimental): Participants in this arm receive a single dose of intravenous tranexamic acid (TXA) during surgery. After skin closure, one breast is treated with topical TXA administered through the surgical drain.
  Interventions: Drug: IV TXA; Drug: Topical TXA
- IV TXA + Topical Saline (Active Comparator): Participants in this arm receive a single dose of intravenous tranexamic acid (TXA) during surgery. After skin closure, one breast is treated with saline administered through the surgical drain.
  Interventions: Drug: IV TXA; Drug: Topical saline
- No IV TXA + Topical TXA (Experimental): Participants in this arm receive no intravenous tranexamic acid (TXA) during surgery. After skin closure, one breast is treated with TXA administered through the surgical drain.
  Interventions: Drug: Topical TXA
- No IV TXA + Topical Saline (Placebo Comparator): Participants in this arm receive no intravenous tranexamic acid (TXA) during surgery. After skin closure, one breast is treated with saline administered through the surgical drain.
  Interventions: Drug: Topical saline

INTERVENTIONS:
Drug: IV TXA — Patients randomized to the IV TXA group will receive intravenous Tranexamic acid during the procedure. The dose will be 1g IV infused over approx. 10 minutes prior to skin closure (dosing of approx. 15 mg/kg, capped at 1 g, which is within safe limits).
  Arms: IV TXA + Topical Saline; IV TXA + Topical TXA
Drug: Topical TXA — Before wound closure, one 15mm round Jackson-Pratt (JP) drain is placed in each breast pocket, exiting through a lateral chest wall stab incision. The randomized topical TXA intervention is then applied through the drain into the breast after skin closure. The drains will then be temporarily clamped for 20 minutes to allow the TXA to dwell in the tissue and exert local effect. After this the clamp is released, the excess fluid sucked off and the drain connected to a drainage bottle.
  Other Names: Topical Tranexamic acid; Topical TXA through drain
  Arms: IV TXA + Topical TXA; No IV TXA + Topical TXA
Drug: Topical saline — Before wound closure, one 15mm round Jackson-Pratt (JP) drain is placed in each breast pocket, exiting through a lateral chest wall stab incision. The randomized saline intervention is then applied through the drain into the breast after skin closure. The drains will then be temporarily clamped for 20 minutes to allow the saline to dwell in the tissue and exert local effect. After this the clamp is released, the excess fluid sucked off and the drain connected to a drainage bottle.
  Other Names: Topical 0.9% Sodium Chloride; Topical Placebo
  Arms: IV TXA + Topical Saline; No IV TXA + Topical Saline

SUMMARY:
This study aims to evaluate whether tranexamic acid (TXA), a medication that helps reduce bleeding, can decrease fluid drainage after breast reduction surgery. Participants will be randomly assigned to receive either intravenous TXA or no TXA during surgery. Additionally, one breast will receive TXA through the surgical drain, while the other will receive saline. This approach allows to compare the effects of TXA on fluid buildup and healing. The goal is to improve recovery and reduce complications after breast reduction surgery.

DETAILED DESCRIPTION:
This single-center, prospective, randomized controlled trial investigates the effect of tranexamic acid (TXA) on postoperative drain output and recovery following bilateral reduction mammaplasty. While TXA is widely utilized to minimize intraoperative blood loss, its role in optimizing postoperative wound healing and fluid management in plastic surgery remains underexplored.

Participants undergoing bilateral breast reduction will be randomized to receive either intravenous TXA or no TXA at the time of surgery. In addition, each breast will be independently randomized to receive TXA or saline via the closed-suction drain after skin closure. This split-body design enables a controlled intra-individual comparison of local TXA effects, while concurrently assessing systemic administration in a parallel fashion.

Primary outcomes include total drain output per breast and time to drain removal. Secondary endpoints include the incidence of postoperative hematoma and patient reported outcomes. All outcome measures will be recorded using standardized protocols and assessed by blinded evaluators where applicable.

Participants will be followed until 30 days postoperatively.

Given the established safety profile of TXA and the relatively low-risk nature of the intervention, no independent data monitoring committee has been appointed. The study has been approved by the local IRB and will adhere to institutional standards for adverse event monitoring and reporting.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Elective bilateral breast reduction
* Patient understands and is willing to participate in the study
* Patient willing to and capable of providing informed consent

Exclusion Criteria:

* Age less than 18 years old
* Prior radiation to the breast
* Secondary/Revision breast reduction
* Known coagulopathy or bleeding disorders
* Intraoperative coagulopathy
* History of seizures
* Active smokers
* Allergy or contraindication to TXA
* Pregnant or breastfeeding patients
* Patient is unable or unwilling to complete the anticipated study follow-up
* Inability to understand the aims and objectives of the study
* Inability to or unwilling to provide informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-11-18 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Total drain output per breast per 24 hours post-surgery (mL) until drain removal | From date of operation until drain removal up to 4 weeks.
  Drain outputs will be recorded separately for each breast twice daily until removal.
Time to drain removal (days) | From date of operation until drain removal up to 4 weeks.
  Drains will be removed per standard protocol by trained staff if the output is ≤30 mL in a 24-hour period for two consecutive days. The time to drain removal will be recorded.

SECONDARY OUTCOMES:
Change in drain fluid color from bloody to serous until drain removal assessed by daily observation | From postoperative Day 1 until drain removal, up to 4 weeks after surgery
  Qualitative change in drain fluid from bloody to serous. Measured by daily observation by clinical staff until drain removal. Change will be recorded as transition from bloody to serous.
Seroma Rate | From date of surgery until end of study (30 days postoperative).
  Rate of clinically evident seromas in the postoperative follow-up period. Diagnosis will be based on physical examination and/or ultrasound when clinically indicated.
Infection Rate | From date of surgery until end of study (30 days postoperative).
  Rate of surgical site infections (superficial or deep) diagnosed based on CDC criteria during the postoperative period.
Hematoma Rate | From date of surgery until end of study (30 days postoperative).
  Rate of postoperative hematoma formation. Diagnosis will be based on physical examination and/or via imaging, if clinically indicated.
Wound Dehiscence Rate | From date of surgery until end of study (30 days postoperative).
  Rate of postoperative wound dehiscence identified clinically, including any spontaneous reopening of the surgical incision.
Length of Hospital Stay | From date of surgery until discharge from the hospital up to 4 weeks.
  Duration of inpatient stay postoperatively, measured in days from the date of surgery to the date of discharge.
30-Day Readmission Rate | From date of surgery until end of study (30 days postoperative)
  Rate of patients readmitted to the hospital within 30 days of the index surgery, regardless of cause.
30-Day Revision Rate | From date of surgery until end of study (30 days postoperative).
  Rate of reoperation or revision procedures performed within 30 days postoperatively due to complications.
Patient-Reported Outcomes (BREAST-Q Breast Reduction Module) | Preoperative before surgery, 7 days after and 30 days after surgery.
  The BREAST-Q Breast Reduction Module is a validated patient-reported outcome measure assessing satisfaction and quality of life following breast reduction surgery. Each subscale is scored from 0 to 100, with higher scores indicating greater satisfaction and/or better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
The investigators do not plan to share individual participant data (IPD) due to institutional and ethical constraints. The informed consent documents did not include provisions for external data sharing, and the dataset contains sensitive clinical information that could pose a risk of re-identification, despite de-identification efforts.

REFERENCES:
- [Background] Nichols G, Andrade E, Gregoski M, Herrera FA, Armstrong MB. Local Infiltration of Tranexamic Acid in Breast Reduction for Symptomatic Macromastia. Ann Plast Surg. 2023 Jun 1;90(6S Suppl 4):S366-S370. doi: 10.1097/SAP.0000000000003456. Epub 2023 Feb 18. PMID 36856723
- [Background] Ausen K, Fossmark R, Spigset O, Pleym H. Randomized clinical trial of topical tranexamic acid after reduction mammoplasty. Br J Surg. 2015 Oct;102(11):1348-53. doi: 10.1002/bjs.9878. PMID 26349843
- [Background] Safran T, Vorstenbosch J, Viezel-Mathieu A, Davison P, Dionisopoulos T. Topical Tranexamic Acid in Breast Reconstruction: A Double-Blind Randomized Controlled Trial. Plast Reconstr Surg. 2023 Oct 1;152(4):699-706. doi: 10.1097/PRS.0000000000010322. Epub 2023 Feb 27. PMID 36827482
- [Background] Liechti R, van de Wall BJM, Hug U, Fritsche E, Franchi A. Tranexamic Acid Use in Breast Surgery: A Systematic Review and Meta-Analysis. Plast Reconstr Surg. 2023 May 1;151(5):949-957. doi: 10.1097/PRS.0000000000010071. Epub 2022 Dec 19. PMID 36729428
- [Background] Guggenheim L, Magni S, Catic A, Pagnamenta A, Harder Y, Schmauss D. The Effects of Systemic Tranexamic Acid Administration on Drainage Volume, Duration of Drain Placement, and Length of Hospital Stay in Skin- and Nipple-Sparing Mastectomies with Immediate Expander-Based Breast Reconstruction. J Clin Med. 2024 Oct 30;13(21):6507. doi: 10.3390/jcm13216507. PMID 39518646
- [Background] Zucal I, De Pellegrin L, Pagnamenta A, Schmauss D, Brucato D, De Monti M, Schweizer R, Harder Y, Parodi C. Topical Application of Tranexamic Acid in Abdominoplasties Leads to Lower Drainage Volume and Earlier Drain Removal. Plast Reconstr Surg Glob Open. 2025 May 20;13(5):e6799. doi: 10.1097/GOX.0000000000006799. eCollection 2025 May. PMID 40395663
- [Background] Fung E, Godek M, Roth JM, Montalmant KE, Yu BZ, Henderson PW. The current state of tranexamic acid in mastectomy and breast reconstruction: A systematic review and meta-analysis. J Plast Reconstr Aesthet Surg. 2025 May;104:259-272. doi: 10.1016/j.bjps.2025.03.022. Epub 2025 Mar 12. PMID 40156946
- [Background] Om A, Marxen T, Kebede S, Losken A. The Usage of Intravenous Tranexamic Acid in Reduction Mammaplasty Safely Reduces Hematoma Rates. Ann Plast Surg. 2023 Jun 1;90(6S Suppl 4):S371-S374. doi: 10.1097/SAP.0000000000003296. Epub 2022 Dec 8. PMID 36729851
- [Background] Buheiri AR, Tveskov L, Dines LM, Bagge JD, Moller S, Bille C. Tranexamic Acid in Breast Surgery - A Systematic Review and Meta-Analysis. Clin Breast Cancer. 2025 Jul;25(5):e496-e510. doi: 10.1016/j.clbc.2025.01.011. Epub 2025 Jan 23. PMID 39924382
- [Background] Ker K, Edwards P, Perel P, Shakur H, Roberts I. Effect of tranexamic acid on surgical bleeding: systematic review and cumulative meta-analysis. BMJ. 2012 May 17;344:e3054. doi: 10.1136/bmj.e3054. PMID 22611164
- [Background] Dunn CJ, Goa KL. Tranexamic acid: a review of its use in surgery and other indications. Drugs. 1999 Jun;57(6):1005-32. doi: 10.2165/00003495-199957060-00017. PMID 10400410
- [Background] Kaoutzanis C, Winocour J, Gupta V, Ganesh Kumar N, Sarosiek K, Wormer B, Tokin C, Grotting JC, Higdon KK. Incidence and Risk Factors for Major Hematomas in Aesthetic Surgery: Analysis of 129,007 Patients. Aesthet Surg J. 2017 Oct 16;37(10):1175-1185. doi: 10.1093/asj/sjx062. PMID 28398469
- [Background] Yao A, Yi J, Greige N, Chemakin K, Weichman KE, Ricci JA. Effect of intraoperative blood pressure on incidence of hematoma in breast reduction mammoplasty. J Plast Reconstr Aesthet Surg. 2022 Aug;75(8):2594-2600. doi: 10.1016/j.bjps.2022.04.014. Epub 2022 Apr 22. PMID 35568688
- [Background] Alhebshi ZA, Sabbagh SR, AlQurain ZJ, Bamuqabel AO, Dahlan DJ, Rajoub RA, Fallatah DO, Rajoub BA, Wasaya HMI, Fallatah E. The Role of Tranexamic Acid Use in Reduction Mammaplasty: A Systematic Review and Meta-Analysis. Aesthet Surg J Open Forum. 2025 May 3;7:ojaf035. doi: 10.1093/asjof/ojaf035. eCollection 2025. PMID 40575008